CLINICAL TRIAL: NCT05854992
Title: Treatments of Migraine with Triptans in Individuals with Elevated Cardiovascular Risk and in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, M. Hassan Murad, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 22-005920
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Migraine; Cardiovascular Diseases; Pregnancy
MeSH Terms: conditions — Migraine Disorders; Cardiovascular Diseases | interventions — Tryptamines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cardiovascular Risk Group Treated with Triptans: Subjects with diagnosis of migraine and cardiovascular disease, cerebrovascular disease and/or two or more cardiovascular risk factors who received Triptans as part of clinical care.
  Interventions: Drug: Acute migraine treatment with any prescribed triptans
- Cardiovascular Risk Control Group Treated with No Triptans: Subjects with who did not received Triptans as part of clinical care.
  Interventions: Drug: Standard of care management of acute migraine without triptans
- Pregnant Women Group Treated with Triptans: Subjects diagnosed with migraine that received Triptans as part of clinical care during pregnancy.
  Interventions: Drug: Acute migraine treatment with any prescribed triptans
- Pregnant Women Control Group Treated with No Triptans: Subjects that did not receive Triptans as part of clinical care during pregnancy.
  Interventions: Drug: Standard of care management of acute migraine without triptans

INTERVENTIONS:
Drug: Acute migraine treatment with any prescribed triptans — Sumatriptan, treximet (sumatriptan/naproxen combination), zolmitriptan, naratriptan, rizatriptan, almotriptan, eletriptan, and frovatriptan. No restriction on dose, frequency, duration, or delivery routes.
  Other Names: Triptans
  Groups: Cardiovascular Risk Group Treated with Triptans; Pregnant Women Group Treated with Triptans
Drug: Standard of care management of acute migraine without triptans — Any standard of care management without triptans
  Other Names: No triptans
  Groups: Cardiovascular Risk Control Group Treated with No Triptans; Pregnant Women Control Group Treated with No Triptans

SUMMARY:
Researchers are evaluating the safety of triptan treatment of migraine in individuals with elevated cardiovascular risk and in pregnant women.

DETAILED DESCRIPTION:
Migraine is a very common condition that can be associated with significant morbidity. For the acute treatment of migraine attacks, the use of triptans, NSAIDs, acetaminophen, dihydroergotamine, calcitonin gene-related peptide antagonists, lasmiditan, and some nonpharmacologic treatments are associated with improved pain and function. The effectiveness of these therapies has been documented in various studies and summarized in systematic reviews. However, systematic reviews have demonstrated evidence gaps in two groups of patients that were excluded from treatment trials. These are patients with cardiovascular disease or at high risk of cardiovascular events, and pregnant women.

Triptans, the mainstay treatment for migraine attacks and the one supported by the highest quality evidence, are considered vasoactive and are contraindicated per formulary in individuals who have a history of myocardial infarction, stroke, or uncontrolled vascular risk factors such as hypertension. These individuals are usually excluded from randomized trials. Similarly, pregnant women have been excluded from triptans trials and the observational studies offered low certainty evidence about their safety. Yet, 44% of surveyed members of the American Headache Society reported being somewhat or very comfortable using triptans in pregnancy.

Therefore, the investigators intend to evaluate the safety of triptan treatment of migraine in individuals with cardiovascular disease or multiple cardiovascular risk factors, and in pregnant women in two target trial emulations.

ELIGIBILITY:
Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk:

Inclusion:

* Aged >=18 years
* At least 1 year history of migraine with or without aura
* Confirmed cardiovascular or cerebrovascular disease, including myocardial infarction (MI), coronary artery disease (CAD), cerebrovascular disease, stroke; or at least 2 cardiovascular risk factors, including diabetes, hyperlipidemia, hypertension, obstructive sleep apnea, peripheral vascular disease;
* At least 1 year of prior triptan treatment or no previous triptan treatment.

Exclusion:

• Prescription of ergot alkaloids or dihydroergotamine within 60 days before or after starting treatment

Treatments of Migraine With Triptans in Pregnant Women

Inclusion:

* Aged >=18 years
* Pregnant woman
* Diagnosis of episodic or chronic migraine with or without aura before pregnancy

Exclusion:

• Prescription of ergot alkaloids or dihydroergotamine <= 60 days before pregnancy or during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were identified through Mayo Clinic electronic health records.
Sampling Method: Non-Probability Sample
Enrollment: 68419 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: number of subjects to experience major adverse cardiovascular events (MACE) which consists of all-cause death, nonfatal myocardial infarction, nonfatal stroke, heart failure, transient cerebral ischemia, or revascularization
Full term birth | 39 0/7 weeks of gestation through 40 6/7 weeks of gestation
  Treatments of Migraine With Triptans in Pregnant Women: number of pregnant women to have a full term birth

SECONDARY OUTCOMES:
all-cause death | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: all-cause death
Nonfatal myocardial infarction | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: nonfatal myocardial infarction
Nonfatal stroke | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: nonfatal stroke
Heart failure | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: Heart failure
Transient cerebral ischemia | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: transient cerebral ischemia
Revascularization | 60 days of starting treatment
  Treatments of Migraine With Triptans in Individuals With Elevated Cardiovascular Risk: revascularization
Pre-term delivery | 37 0/7 weeks of gestation through 38 6/7 weeks of gestation
  Treatments of Migraine With Triptans in Pregnant Women: Pre-term delivery
Cesarean section delivery | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: cesarean section delivery
Spontaneous abortions/miscarriage | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Spontaneous abortions/miscarriage
Fetal death/stillbirth | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Fetal death/stillbirth
Intra-uterine growth restriction | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Intra-uterine growth restriction
Eclampsia/preeclampsia | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Eclampsia/preeclampsia
Tubal or ectopic pregnancy | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Tubal or ectopic pregnancy
Major fetal malformations | up to delivery
  Treatments of Migraine With Triptans in Pregnant Women: Major fetal malformations

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Murad, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, VanderPluym JH, Halker Singh RB, Alsibai RA, Roellinger DL, Murad MH. Safety of Triptans in Treating Migraines in Pregnant Women: A Target Trial Emulation. Mayo Clin Proc. 2025 Nov;100(11):1956-1962. doi: 10.1016/j.mayocp.2025.01.023. Epub 2025 Jul 28. PMID 40719668
- [Derived] Wang Z, VanderPluym JH, Halker Singh RB, Alsibai RA, Roellinger DL, Firwana M, Murad MH. Safety of Triptans in Patients Who Have or Are at High Risk for Cardiovascular Disease: A Target Trial Emulation. Mayo Clin Proc. 2024 Nov;99(11):1722-1731. doi: 10.1016/j.mayocp.2024.03.023. Epub 2024 Aug 30. PMID 39207344
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials